CLINICAL TRIAL: NCT01029574
Title: Platelet Rich Plasma on Arthroscopic Repair of the Complete Rotator Cuff Lesions: a Prospective and Randomized Study
Brief Title: Platelet Rich Plasma on Rotator Cuff Repair
Acronym: PRP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Criogenesis (Unknown)
Responsible Party: Principal Investigator, Eduardo Angeli Malavolta, Dr, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0292/08
Record Dates: First submitted 2009-12-09; First posted 2009-12-10 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Rotator Cuff Tears
Keywords: Rotator cuff lesions; Platelet rich plasma; Arthroscopic repair
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rotator cuff repair plus PRP (Experimental): Conventional arthroscopic repair of rotator cuff with application of PRP.
  Interventions: Other: Platelet rich plasma
- Rotator cuff repair alone (Placebo Comparator): Conventional arthroscopic repair of rotator cuff without application of PRP
  Interventions: Other: Platelet rich plasma

INTERVENTIONS:
Other: Platelet rich plasma — Ultra-centrifuged PRP, 40ml, in the liquid way, after portal closure.

SUMMARY:
Repair of the rotator cuff has high rates of re-rupture (20-54%), despite good clinical results. Several ways to improve the healing tendon-bone are currently studied, among them the most used is the use of growth factors. The platelet-rich plasma is a source of several growth factors, and is already used in various orthopedic procedures. The aim of this study is to evaluate the effectiveness of platelet-rich plasma in improve tendon-bone healing in arthroscopic rotator cuff repairs.

DETAILED DESCRIPTION:
Rotator cuff repair(RCR) is a procedure widely performed in the shoulder surgery, given the high prevalence of this type of injury in the population. Regardless of the approach employed, the procedure consists of the rehabilitation of the rotator cuff to his bed. Despite the clinical results are highly satisfactory (success rate around 85%), studies using ultrasound and magnetic resonance imaging (MRI) showed a rate of re-rupture after surgery 20 to 54%. These levels of re-injury suggest a sub-optimal healing in the bone-tendon interface.

Attempts to improve the healing in place of the RMR has been extensively studied in the orthopedic literature. One is the use of growth factors (GF), cytokines play an important role in chemotaxis, cell proliferation and differentiation, as well as the synthesis of extracellular matrix, and that theoretically could have beneficial role in tissue repair.

The Platelet-Rich Plasma (PRP) is one of the most studied sources of GF. It is easy to prepare and non-immunogenic (is done with the patient's own blood), and has the further advantage of the presence of several FC (including PDGF, bFGF, TGF-B, VEGF, EGF, CTGF and IGF). This fact is important because the disease have different effects on different receivers during the various stages of healing.

The use of PRP in bone healing has been evaluated in several studies with conflicting results. There are preclinical studies demonstrating the beneficial effect of PRP on tendon and ligament repair. However, there is no published papers showing the effectiveness of the use of PRP on tendon-bone interface.

The aim of this study is to evaluate the effectiveness of PRP in enhancing the healing tendon-bone repair after injury of RC.

Will be operated patients with complete injury (full thickness) of the rotator cuff, divided into two groups randomly. The use of PRP or not will be decided by sealed envelopes, with 20 individuals in each group. The subjects will be assessed pre and postoperatively according to the criteria for the Constant and UCLA and with the help of MRI, being unknown to the evaluators to which group the patient belongs.

ELIGIBILITY:
Inclusion Criteria:

* Pain or functional deficit in the shoulder to justify surgical intervention;
* Complete lesion(full thickness) of the supraspinatus tendon resulting from trauma or degenerative confirmed by MRI;
* Patients skeletally mature, regardless of sex;
* Signing the consent form.

Exclusion Criteria:

* Psychiatric disorders;
* Vascular-nerve lesions affecting the upper limb;
* Pregnancy;
* Immature skeleton;
* Comorbidities unmatched clinically;
* Osteoarthritis of the acromioclavicular joint symptomatic requiring surgical intervention;
* Glenohumeral arthrosis grades 2, 3 and 4 Samilson and Prieto;
* Rotator Cuff Arthropathy grades IB, IIA and IIB of Seebauer;
* Active or recent infection;
* Neuropathic arthropathy;
* Previous surgery on the same shoulder operated;
* Patients with painful pathologies of the cervical spine;
* Patients diagnosed with fibromyalgia;
* Patients who do not understand or do not agree with the consent form;
* Fatty degeneration of the muscles of the MR resonance;
* Retraction of the tendon greater than 3cm (MRI or intraoperative);
* Subscapular or Infraspinatus rupture that needs repair (MRI or intraoperative).

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
UCLA Score | 12 months

SECONDARY OUTCOMES:
Constant Scores and Re-tear rate (MRI) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo A Malavolta, MD, Principal Investigator — University of Sao Paulo - Orthopedic and Traumatology Department; Arnaldo A Ferreira Neto, PhD, Study Director — University of Sao Paulo - Orthopedic and Traumatology Department
Locations (2):
- Brazil (2):
  - University of São Paulo - Orthopedics and traumatology department, São Paulo, São Paulo
  - University of São Paulo, São Paulo, São Paulo

REFERENCES:
- [Derived] Malavolta EA, Gracitelli MEC, Assuncao JH, Ferreira Neto AA, Bordalo-Rodrigues M, de Camargo OP. Clinical and Structural Evaluations of Rotator Cuff Repair With and Without Added Platelet-Rich Plasma at 5-Year Follow-up: A Prospective Randomized Study. Am J Sports Med. 2018 Nov;46(13):3134-3141. doi: 10.1177/0363546518795895. Epub 2018 Sep 20. PMID 30234999